CLINICAL TRIAL: NCT05589610
Title: An Open-label, Phase 2 Study to Assess the Safety and Efficacy of EQ101 in Adult Subjects With Moderate to Severe Alopecia Areata
Brief Title: Study of EQ101 in Adult Subjects With Moderate to Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Equillium (Industry)
Collaborators: Equillium AUS Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQ101-104-01
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Alopecia Areata; Alopecia; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EQ101 (Experimental): EQ101 weekly
  Interventions: Drug: EQ101

INTERVENTIONS:
Drug: EQ101 — EQ101, 2 mg/kg, once weekly dosing, for a total of 24 doses

SUMMARY:
The purpose of this study is to assess the safety, PK, and PD of EQ101 as well as measure the efficacy of EQ101 at Week 24 compared to Baseline in adult subjects with moderate to severe AA. The study consists of 3 phases: a screening phase of up to 5 weeks, a treatment phase of 24 weeks, and a follow-up phase of 4 weeks. Study drug will be administered via intravenous (IV) push weekly.

DETAILED DESCRIPTION:
This is a multicentre, Phase 2, open-label PoC study of EQ101 in adult subjects with at least 35% scalp hair loss due to AA. Approximately, 30 subjects will be enrolled in the study. During the 24-week treatment period, subjects will be dosed once weekly with EQ101 2 mg/kg IV. Subjects then will be followed up for an additional 4 weeks. The maximum duration of study participation will be approximately 33 weeks.

Eligible subjects must be between the ages of 18 and 60 years, have a clinical diagnosis of AA with a scalp hair loss of ≥ 35% at Screening and Baseline. Approximately 25% of subjects with 35% to < 50% scalp hair loss and approximately 25% may have AT and/or AU. In addition, each subject's current hair loss episode must have lasted at least 6 months but not more than 7 years and there can be no appreciable improvement in terminal hair regrowth within 6 months of Baseline.

Safety, efficacy, PK, and PD assessments will be made during the study. Safety assessments will include AEs (i.e., type, severity, frequency, seriousness, causality) and clinical safety lab results. Efficacy measurements will include Clinical Investigator assessments (e.g., SALT, ClinRO for eyebrows (EB), eyelashes (EL), and body hair changes) and assessments made by study subjects (e.g., Scalp Hair Assessment PRO, and PRO measures for EB, EL, and body hair changes).

ELIGIBILITY:
Key Inclusion Criteria:

1.Subjects have AA, meeting all of the following criteria:

1. Clinical diagnosis of AA with no other aetiology of hair loss ;
2. At least 35% scalp hair loss, as defined by a SALT score ≥ 35, at Screening and Baseline. Approximately 25% of subjects with 35% to <50% scalp hair loss and 25% may have AT/AU.
3. Current episode of hair loss lasting > 6 months to < 7 yrs at time of Screening; and
4. No appreciable change in terminal hair regrowth within 6 months of the baseline visit.

Key Exclusion Criteria:

1. Known history of, or currently experiencing, male pattern androgenetic alopecia or female pattern hair loss
2. History of scalp hair transplantation.
3. Other scalp disease that may impact AA assessment or require topical treatment
4. Unwilling to maintain a consistent hair style, including shampoo and hair products, and to refrain from weaves or extensions throughout the course of the study, or shaving of scalp.
5. Use of adhesive or difficult to remove hairpiece or wigs during the study
6. Have undergone significant trauma or major surgery within 8 weeks of the first dose of study drug or considered in imminent need for surgery or with elective surgery scheduled to occur during the study.
7. Participation in other clinical studies involving investigational drug(s) within 4 weeks prior to the baseline visit.
8. Treatment with an oral JAK inhibitor within 6 months prior to the baseline visit.
9. Have previously been treated with an oral JAK inhibitor for AA for at least 12 weeks without achieving at least a 25% improvement in SALT score.
10. Have been treated with any cell-depleting agents including but not limited to rituximab: within 6 months of the baseline visit, or 5 half-lives (if known), or until lymphocyte count returns to normal, whichever is longer.
11. Have been treated with any biologics within 12 weeks or 5 half-lives of the baseline visit, whichever is longer.
12. Have been treated with any oral immune suppressants within 8 weeks of the baseline visit.
13. Have received intralesional injections of corticosteroid or platelet-rich plasma (PRP) in the scalp within 6 weeks of the baseline visit.
14. Have used phototherapy, contact sensitisers, contact irritants, or cryotherapy within 4 weeks of the baseline visit.
15. Have used topical treatments applied to the scalp, eyebrows, or eyelashes (e.g., corticosteroid cream; JAK inhibitors; medicated shampoo; minoxidil (Rogaine); or herbal hair care that could affect AA) within 4 weeks of the baseline visit.
16. Have current or recent history of clinically significant severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality
17. Have a known immunodeficiency disorder.
18. History of solid organ or haematological transplantation.
19. History of a lymphoproliferative disease or malignancy, other than adequately treated non-melanoma skin cancer or cervical carcinoma with no evidence of recurrence.
20. Have active acute or chronic infection
21. Abnormalities in clinical laboratory tests at Screening:

    1. Absolute neutrophil count (ANC) <1.0 × 109/L.
    2. Liver function tests ( ALT and AST) >3 x ULN.
    3. Total bilirubin >1.5 times ULN (unless isolated Gilbert's syndrome)
    4. Serum creatinine >1.5 ULN.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Sinclair Dermatology, East Melbourne
  - Fremantle Dermatology, Fremantle
  - Premier Specialists, Kogarah
  - Veracity Clinical Research, Woolloongabba
- Optimal Clinical Trials Limited, Auckland, New Zealand

REFERENCES:
- See also: Company website — https://www.equilliumbio.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EQ101
Started | 36
Completed | 30
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | EQ101
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 12
  Australia | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Week 28
Measure: Count of Participants; unit: Participants
Arm/Group | EQ101
Number analyzed (Participants) | 36
Participants | 27

2. Secondary Outcome: The Efficacy of EQ101 in Adult Subjects With Moderate to Severe Alopecia
Description: Percent change in SALT score
Time Frame: Week 24
Reporting Status: Not Posted

3. Secondary Outcome: To Characterize the Pharmacokinetics (PK) of EQ101
Description: To characterize the pharmacokinetics (PK) of EQ101 by plasma concentrations
Time Frame: Week 24
Reporting Status: Not Posted

4. Secondary Outcome: To Characterize the Pharmacodynamics (PD) of EQ101
Description: Percent change in target engagement
Time Frame: Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing the ICF through week 28 (final follow-up visit) for a total of approximately 33 weeks (5 week screening period starting with the signing of the ICF, 24 week treatment period, and 4 week follow up period), all SAEs and nonserious AEs will be recorded on the SAE/AE eCRF.
Arm/Group | EQ101
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 11/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ101 (N=36)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Fatigue (General disorders) | 4 (26)
Headache (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT05589610/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT05589610/SAP_001.pdf